CLINICAL TRIAL: NCT01912560
Title: A Randomized, Double-Blind, Placebo-Controlled Pilot Study to Assess the Safety, Efficacy and Pharmacodynamics of CAT-2003 Alone and In Combination With A Statin in Patients With Hyperlipidemia (PATHWAYS I)
Brief Title: Pilot Study To Assess CAT-2003 in Patients With Hyperlipidemia
Acronym: PATHWAYS I
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Catabasis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAT-2003-201
Record Dates: First submitted 2013-07-25; First posted 2013-07-31 (Estimated); Last update posted 2016-07-28 (Estimated); Status verified 2016-07

CONDITIONS: Dyslipidemia; Hypercholesterolemia; Hypertriglyceridemia
MeSH Terms: conditions — Dyslipidemias; Hypercholesterolemia; Hypertriglyceridemia | interventions — Hydroxymethylglutaryl-CoA Reductase Inhibitors

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- CAT-2003 or Placebo Dose 1 (Experimental): Daily for 28 days in patients with moderate hypertriglyceridemia
  Interventions: Drug: CAT-2003; Drug: Placebo
- CAT-2003 or Placebo Dose 2 (Experimental): Daily for 28 days in patients with moderate hypertriglyceridemia
  Interventions: Drug: CAT-2003; Drug: Placebo
- CAT-2003 or Placebo Dose 3 (Experimental): Daily for 28 days in patients with moderate hypertriglyceridemia
  Interventions: Drug: CAT-2003; Drug: Placebo
- CAT-2003 or Placebo Dose 4 (Experimental): Daily for 28 days in patients with hypercholesterolemia who are on a statin
  Interventions: Drug: CAT-2003; Drug: Placebo; Drug: Statin

INTERVENTIONS:
Drug: CAT-2003
Drug: Placebo
Drug: Statin — All patients being treated with a stable dose of a statin prior to enrollment continue on their dosing regimen.
  Arms: CAT-2003 or Placebo Dose 4

SUMMARY:
The purpose of this study is to determine the safety and efficacy of different doses of CAT-2003 in patients with hyperlipidemia when CAT-2003 is taken for 4 weeks. The study will evaluate effects of CAT-2003 on (1) fasting triglycerides and non-HDL-C in patients with moderate hypertriglyceridemia and (2) fasting LDL-C levels in combination with a statin in patients with hypercholesterolemia who are on a statin.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 69 years at Screening
* Hypertriglyceridemia (TG ≥ 200 mg/dL and < 500 mg/dL and non-HDL-C ≥ 100 mg/dL and < 220 mg/dL) OR
* Hypercholesterolemia (LDL-C ≥ 100 mg/dL and < 190 mg/dL and TG value < 200 mg/dL) plus a stable dose of statin for at least 4 weeks prior to Screening.
* Body mass index (BMI) ≤ 45 kg/m2

Exclusion Criteria:

* History of any major cardiovascular event within 6 months of Screening
* Type I diabetes mellitus
* Any condition that may predispose the patient to secondary hyperlipidemia, such as uncontrolled hypothyroidism
* Any statin at the highest approved dose
* Non-statin lipid-altering drugs other than cholesterol absorption inhibitors.
* Active peptic ulcer disease or a history of muscle disease or myopathy

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2013-07; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Absolute and percent change from baseline in plasma triglycerides in patients with hypertriglyceridemia | 4 weeks
Absolute and percent change from baseline in plasma low density lipoprotein-cholesterol in patients with hypercholesterolemia | 4 weeks

SECONDARY OUTCOMES:
Absolute and percent change from baseline in plasma non-high-density lipoprotein cholesterol | 4 weeks
Pharmacodynamic effects of CAT-2003 on other lipid biomarkers in patients with hyperlipidemia | 4 weeks
Frequency of adverse events | 4 weeks
  Safety and tolerability will be assessed for all enrolled patients from the time the patient signs the informed consent through post-treatment follow-up. Safety parameters include physical exam, vital signs, clinical laboratory tests, ECGs and concomitant medications.

CONTACTS AND LOCATIONS:
Locations (11):
- United States (10):
  - Muscle Shoals, Alabama
  - Los Angeles, California
  - Jacksonville, Florida
  - Miami, Florida
  - Winter Park, Florida
  - Kansas City, Kansas
  - Louisville, Kentucky
  - Auburn, Maine
  - Raleigh, North Carolina
  - Cincinnati, Ohio
- Sainte-Foy, Quebec, Canada